CLINICAL TRIAL: NCT01481818
Title: Phase Ⅰ,ⅡStudy of Topically Applied Green Tea Extract for Prevention and Treatment of Radio Dermatitis and Radiation Mucositis
Brief Title: Study of Topically Applied Green Tea Extract for Radio Dermatitis and Radiation Mucositis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Han Xi Zhao, M.D., Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GTERD2011
Record Dates: First submitted 2011-11-23; First posted 2011-11-30 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Epigallocatechin Gallate; Radio Dermatitis; Radiation Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- radioprotector (Experimental)
  Interventions: Drug: EGCG

INTERVENTIONS:
Drug: EGCG — Apply about 0.05ml/cm2 EGCG with different concentration topically for 3 times a day during radiotherapy

SUMMARY:
Radiodermatitis and radiation mucositis were the most frequent side-effect during the course of radiotherapy, especially when concurrent chemoradiotherapy applied. Since reactive oxygen species formed upon radiation therapy play a central role in initiating and driving the detrimental signaling events, antioxidant supplementation is thought to provide a photoprotective effect against radiation. Green tea extract has been shown to have antioxidant and anti-inflammatory effects on various types of cells. To evaluate the safety and efficiency of green tea extract in the treatment of radio dermatitis and radiation mucositis, the investigators conducted this phase Ⅰ,II study using topical EGCG in cancer patients receiving radiotherapy or concurrent chemoradiotherapy .

DETAILED DESCRIPTION:
The phase 1 trial using EGCG for prevention and treatment radiodermatitis in patients with breast cancer.

Patient selection criteria The eligible criteria including: ≥18 years old; adequate renal and hepatic function; with histological proven breast cancer; receive adjuvant external electron beam RT to chest wall (with or without lymph nodes associated) after modified radical mastectomy; receive at least 50.0 Gy in 25~28 fractions, delivered daily, 5d/week; each treatment was planned using a simulated locator with the patient in the supine position and adequate immobilization.

The exclusion criteria were as follows: previous RT to chest wall and/or lymph nodes associated; previous chemotherapy or radiotherapy for another neoplasia; pregnancy or lactation; concomitant chemotherapy; a known allergy or hypersensitivity to EGCG.

Treatment Protocol Patients were instructed to apply about 0.01~0.05ml/cm2 EGCG 3 times a day to the area under treatment. The initial concentration is about 40μM, adjusted from previous study (Katiyar SK, Afaq F, Perez A, Mukhtar H. Green tea polyphenol (-)-epigallocatechin-3-gallate treatment of human skin inhibits ultraviolet radiation-induced oxidative stress. Carcinogenesis. 2001; 22(2):287-94) EGCG treatment begins when cutaneous toxicity reaches grade 1, evaluated by the principal investigator and the patient's radiation oncologist according to Radiation Therapy Oncology Group acute skin toxicity scale.The duration of EGCG treatment will last at least two weeks after RT completion, further use of EGCG was not encouraged.

At per protocol, patients who developed grade Ⅱ radiation-induced dermatitis had the option to either withdraw from the study or to continue with EGCG.Adverse events more than grade 1 attributed to EGCG that did not respond to supportive care were considered dose-limiting toxicity (DLT). Transient toxicity more than grade 1 that responded to supportive care was recorded as an adverse event but was not considered dose limiting. In general, for grade 2 adverse events attributed to EGCG, therapy was held until symptoms resolved to ≤ grade 1 and then reinitiated along with supportive care measures at the same dose level. The maximum-tolerated dose (MTD) was defined as the dose level below the lowest dose that induced a DLT in at least one third of patients (at least two of six patients) after one cycle of therapy.

Acute skin toxicity were evaluated using Radiation Therapy Oncology Group acute skin toxicity scale by principal investigator. The Skin Toxicity Assessment Tool was used to measure patient-reported discomforts. (Berthelet E, Truong PT, Musso K, et al. Preliminary reliability and validity testing of a new Skin Toxicity Assessment Tool (STAT) in breast cancer patients undergoing radiotherapy. Am J Clin Oncol 2004;27:626-631.).

Statistical Analyses The primary outcome for this phase I trial was the number of DLTs and determination of the MTD, with frequency and severity of radiodermatitis the secondary outcome, frequency and severity of pain and pruritus the third outcome.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* with histologically proven cancer
* receive external radiotherapy or concurrent chemoradiotherapy

Exclusion Criteria:

* previous radiotherapy
* previous chemotherapy for another neoplasia
* pregnancy or lactation
* a known allergy or hypersensitivity to EGCG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-09; Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | participants will be followed for the duration of radiotherapy, an expected average of 6 weeks").

SECONDARY OUTCOMES:
Frequency and Severity of Radio Dermatitis or Radiation Mucositis during Radiotherapy | participants will be followed every weeks for the duration of radiotherapy, an expected average of 6 weeks").

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, M.D., Study Director — Shandong Cancer Hospital and Institute

REFERENCES:
- [Derived] Zhao H, Zhu W, Xie P, Li H, Zhang X, Sun X, Yu J, Xing L. A phase I study of concurrent chemotherapy and thoracic radiotherapy with oral epigallocatechin-3-gallate protection in patients with locally advanced stage III non-small-cell lung cancer. Radiother Oncol. 2014 Jan;110(1):132-6. doi: 10.1016/j.radonc.2013.10.014. Epub 2014 Jan 17. PMID 24444526